CLINICAL TRIAL: NCT07095231
Title: A Phase 1 Dose Escalation Study to Assess the Safety, Reactogenicity, and Immunogenicity of STX-S for Prevention of SARS-CoV-2 Infection as a Booster Dose
Brief Title: Safety, Reactogenicity, and Immunogenicity Trial of STX-S SARS-CoV-2 Vaccine in Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 24-1104
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07-17

CONDITIONS: COVID-19
Keywords: Booster Dose; Capricor; coronavirus; Dose-Escalation; NextGen; phase 1; STX-S; vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Healthy adult participants, 18 to 64 years of age, will be administered a single intramuscular dose of STX-S at 25 ng at a volume of 0.25 mL. Three sentinel participants, aged < 50, will be enrolled over at least 2 days. The Protocol Safety Review Team (PSRT) will conduct a safety review before enrolling the remainder of the cohort. N=20
  Interventions: Biological: STX-S
- Cohort 2 (Experimental): Healthy adult participants, 18 to 64 years of age, will be administered a single intramuscular dose of STX-S at 50 ng at a volume of 0.5 mL. N=20
  Interventions: Biological: STX-S
- Cohort 3 (Experimental): Healthy adult participants, 18 to 64 years of age, will be administered a single intramuscular dose of STX-S at 125 ng at a volume of 0.5 mL. N=20
  Interventions: Biological: STX-S

INTERVENTIONS:
Biological: STX-S — A proprietary vaccine developed internally by Capricor utilizing exosomes that were engineered to express spike proteins on the surface

SUMMARY:
This phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of STX-S in adults who have previously received a primary series and at least one booster with an authorized or licensed SARS-CoV-2 parenteral vaccine. The study is designed as a non-randomized, open-label, dose-escalation clinical trial evaluating three dose levels of STX-S. A sample size of 60 participants (20 participants per dose cohort) is anticipated. The primary objective is to evaluate the safety and reactogenicity of a single intramuscular (IM) injection of three different dose levels (25 ng, 50 ng, and 125 ng) of STX-S in previously vaccinated healthy adults.

DETAILED DESCRIPTION:
This phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of STX-S in adults who have previously received a primary series and at least one booster with an authorized or licensed SARS-CoV-2 parenteral vaccine. The study is designed as a non-randomized, open-label, dose-escalation clinical trial evaluating three dose levels of STX-S. A sample size of 60 participants (20 participants per dose cohort) is anticipated. The primary objective is to evaluate the safety and reactogenicity of a single intramuscular injection of three different dose levels (25 ng, 50 ng, and 125 ng) of STX-S in previously vaccinated healthy adults. The secondary objectives are to evaluate the systemic anti-Spike humoral immune responses of a single Intramuscular (IM) injection of STX-S and to evaluate nasal mucosal Immunoglobulin A (IgA) and Immunoglobulin G (IgG) responses after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent before initiation of any study procedures.
2. Able to understand and agree to comply with planned study procedures and be available for all study visits.
3. Non-pregnant adults, 18 through 64 years of age at the time of vaccination.
4. Participants of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception***

   *These criteria apply to females who are in a heterosexual relationship who are of childbearing potential. Not of childbearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation/salpingectomy).

   **True abstinence is 100% of the time, no sexual intercourse (penis enters the vagina). Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods.

   ***Acceptable forms of primary contraception include a monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more before the participant's vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable/transdermal hormonal birth control products. Must have used at least one acceptable primary form of contraception for at least 30 days before vaccination and agree to continue at least one acceptable primary form of contraception through 60 days after vaccination.
5. Male participants must use acceptable contraception* or be vasectomized and must refrain from donating sperm for 60 days following study vaccination.

   *Acceptable contraception includes abstinence from intercourse with a female participant of childbearing potential or use of a male condom. Contraception use does not apply to males in an exclusively same-sex relationship.
6. Participants of childbearing potential must have a negative urine pregnancy test at screening and within 24 hours before study vaccination.
7. In general good health.* *As determined by medical history and physical examination, including vital signs, to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of the safety of participants. Chronic medical diagnoses/ conditions should be stable for the last 30 days (i.e., no hospitalizations, emergency room (ER), or urgent care for the condition). This includes no change in chronic prescription medication, dose, or frequency due to deterioration of the chronic medical diagnosis/condition 30 days before the study vaccination. Any prescription change, due to a change of health care provider, insurance company, etc., or done for financial reasons and in the same class of medication will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as-needed (prn) medications if, in the opinion of the participating site Principal Investigator or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity.
8. Receipt of a complete primary authorized or approved COVID-19 vaccine series and at least one booster* with the last vaccination at least 16 weeks before study vaccination.

   *Booster may be either homologous or heterologous to the primary vaccine series. It must be a Food and Drug Administration (FDA)-authorized/licensed vaccine, though doses may have been received during a clinical trial.
9. Clinical screening laboratory evaluations are within normal reference ranges or grade 1 with no clinical significance (NCS) per the investigator's discretion.* *(White Blood Cells [WBCs] with differential, hemoglobin [Hgb], platelets [PLTs], Alanine Transaminase [ALT], Aspartate Transaminase [AST], Creatinine [Cr], Alkaline Phosphatase [ALP], Total Bilirubin [T. Bili]). ALT, AST, ALP, T. Bili, and creatinine values below the reference range will not be exclusionary as these values below the reference range are clinically insignificant.
10. Must agree to have samples stored for secondary research.

Exclusion Criteria:

1. Positive SARS-CoV-2 PCR at screening.
2. Abnormal vital signs (Grade 1 or higher)*:

   *Grade 1 or higher is equivalent to: Systolic blood pressure (SBP) >/= 141 mmHg or </= 89 mmHg Diastolic blood pressure (DBP) >/= 91 mmHg Heart rate (HR) is >/= 101 beats per minute or </= 54 beats per minute Oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)
3. History of SARS-CoV-2 infection or receipt of any COVID-19 vaccine < 16 weeks prior to study vaccination.
4. Participant who is pregnant or breastfeeding.
5. Blood or plasma donation within 4 weeks before study vaccination.
6. Receipt of antibody or blood-derived products within 90 days before study vaccination.
7. Any self-reported or documented significant medical or psychiatric diseases* or any other condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.

   *Significant medical or psychiatric conditions include but are not limited to significant kidney disease, liver disease, ongoing malignancy, or recent diagnosis of malignancy in the last five years, excluding treated basal and squamous cell carcinoma of the skin and cervical carcinoma in situ, which are allowed.
8. Neurological or neurodevelopmental conditions*

   *Including history of Bell's palsy, history of four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care, epilepsy, seizures in the last 5 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease.
9. History of significant respiratory disease requiring daily medications currently, history of asthma in the past 5 years, or any treatment of respiratory disease exacerbations in the last 5 years.
10. History of cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), including any history of myocarditis, pericarditis, or uncontrolled cardiac arrhythmia.
11. Any autoimmune disease, including hypothyroidism, without a defined non-autoimmune cause.
12. Has an acute illness determined by the site Principal Investigator or appropriate sub-investigator within 72 hours before study vaccination*.

    *An acute illness that is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site Principal Investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
13. Has a positive test result for hepatitis B surface antigen, hepatitis C virus RNA (by reflex testing), or human immunodeficiency virus (HIV) antigen/antibody test at screening.
14. Has any confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections, and chronic* immunosuppressant medication within the past 6 months.**

    *Chronic means more than 14 continuous days.

    **Ophthalmic and topical steroids are allowed. See exclusion 19 for intranasal steroids.
15. Has received any investigational product within 60 days, or 5 half-lives, whichever is longer, before vaccination or is planning to receive one during the study.
16. Has a history of hypersensitivity or severe allergic reaction* to any previous licensed or unlicensed vaccine or the candidate vaccine components.**

    *(e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction)

    **See Investigative Brochure (IB) for vaccine formulation.
17. Received or plans to receive licensed inactivated/subunit vaccine within 14 days of study vaccine administration or live vaccine within 28 days of study vaccine administration.
18. Plan to receive a COVID-19 booster vaccine within the 180 days following study vaccination.
19. Regular use of intranasal medications, including steroids*

    *Participants must have had no intranasal medication use for 30 days before study vaccination and do not plan to use intranasal medications for 30 days after study vaccination for medications other than steroids and for 3 months after study vaccination for intranasal steroids (including over-the-counter (OTC) fluticasone).
20. Use of intranasal illicit drugs in the 5 years before study vaccination or plans to use during the study.
21. Current smoker (including cigarettes, marijuana, and vaping) or smoking within the prior 3 months.
22. Planned international travel between vaccination and Day 29 visit.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of abnormal clinical safety laboratory adverse events (AE). | Through Day 8
Occurrence of adverse events of special interest (AESI) | Through 6 months post-vaccination
Occurrence of medically attended adverse events (MAAEs) | Through 6 months post-vaccination
Occurrence of new onset chronic medical conditions (NOCMCs) | Through 6 months post-vaccination
Occurrence of serious adverse events (SAEs) | Through 6 months post-vaccination
Occurrence of solicited local adverse events (AEs). | Through Day 7 post-vaccination
Occurrence of solicited systemic adverse events (AE). | Through Day 7 post-vaccination
Occurrence of unsolicited adverse events (AE). | Through Day 28 post-vaccination

SECONDARY OUTCOMES:
Nasal mucosal anti-spike binding IgA antibodies | Day 1 through Day 91
Nasal mucosal anti-spike binding IgG antibodies | Day 1 through Day 91
Serum Anti-spike binding Immunoglobulin A (IgA) antibody | Day 1 through Day 181
Serum Anti-spike binding Immunoglobulin G (IgG) antibody | Day 1 through Day 181
Serum Anti-spike neutralizing antibodies | Day 1 through Day 181

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington